CLINICAL TRIAL: NCT04867603
Title: Digital PET/CT Using [Ga-68]PSMA for Characterization of Prostate Lesions
Status: Completed | Type: Observational
Sponsor: Norbert Avril, M.D. (Other)
Responsible Party: Sponsor-Investigator, Norbert Avril, M.D., Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Other Study IDs: CASE1821
Record Dates: First submitted 2021-02-04; First posted 2021-04-30 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Digital PET/CT using [Ga-68]PSMA: Following prostate Standard of Care MRI, eligible participants will receive a single injection of [Ga-68]PSMA followed by digital PET/CT imaging approximately 60 minutes later. PET/CT takes approximately 30-35 minutes, where the participant would lay still on a scanner table.
  Interventions: Drug: [Ga-68]PSMA; Device: PET/CT imaging

INTERVENTIONS:
Drug: [Ga-68]PSMA — The injectable activity will be a maximum of 210 MBq (6.0 mCi) [Ga-68]PSMA at the time of injection and is administered to subjects by intravenous injection.
Device: PET/CT imaging — PET/CT imaging procedure

SUMMARY:
The purpose of this study is to evaluate a radioactive diagnostic study drug, which is called Gallium-68 Prostate Specific Membrane Antigen ([Ga-68]PSMA) for characterization of prostate abnormalities.

DETAILED DESCRIPTION:
Individuals with clinical suspicion of prostate cancer and without prior prostate biopsy are offered abbreviated bi-parametric prostate MRI. As Standard of Care (SOC), MRIs will be examined and scored for likelihood for malignancy using the PI-RADS version 2.1 criteria. Those with PI-RADS 3, 4 or 5 lesions or those with PI-RADS 1 or 2 lesions with clinical suspicion for prostate cancer based on serum PSA level, family history or clinical examination (positive digital rectal examination) will be included on study. Only those receiving care at University Hospitals Cleveland Medical Center will be included into the study.

This study is to evaluate ([Ga-68]PSMA) for characterization of prostate abnormalities. For imaging, an FDA approved imaging technology, digital Positron Emission Tomography (PET/CT) will be used. The study team would like to know if digital PET/CT using [Ga-68]PSMA provides accurate information whether or not a participant has prostate cancer and if there is potential spread of the disease within the body. [Ga-68]PSMA is an investigational (experimental) drug that works by binding to Prostate Specific Membrane Antigen (PSA), which is overexpressed in prostate cancer. [Ga-68]PSMA is experimental because it is not approved by the Food and Drug Administration (FDA). However, FDA approval has been obtained for this study protocol by an Investigational New Drug (IND) application.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a clinical suspicion of prostate cancer defined by PI-RADS 3, 4 or 5 lesions detected on MRI as well as patients with negative prostate MRI or those with PI-RADS 1 or 2 lesions if they have continued suspicion for prostate cancer. Patients who cannot undergo MRI imaging but have a clinical suspicion for prostate cancer based on serum PSA level, family history or clinical examination (positive digital rectal examination) can also be included.
* Able to tolerate PET/CT scans
* Informed consent must be given and signed

Exclusion Criteria:

* Anti-cancer treatment (chemotherapy and/or radiation therapy) within the last 2 weeks
* Known allergy against Ga-68 PSMA
* Prior prostate biopsy within the last 2 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants who are at least 18 years old with a clinical suspicion of prostate cancer. Patients are referred from the Urology Institute within the University Hospitals Health System.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
True positive rate | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by true-positive rate. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
False positive rate | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by false-positive rate. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
True negative rate | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by true negative rate. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
False negative negative rate | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by false negative rate. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
Sensitivity | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by sensitivity. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
Specificity | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by specificity. The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
Positive predictive value (PPV) | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by (PPV). The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
Negative predictive value (NPV) | During scan, up to 35 minutes
  Diagnostic performance of digital PET/CT using [Ga-68]PSMA for characterization of prostate lesions, as measured by (NPV). The uptake of [Ga-68]PSMA within the prostate gland will be visually assessed and compared to surrounding tracer uptake within the prostate gland. The majority of participants will subsequently undergo prostate biopsy as part of routine clinical work-up. Subsequent histopathology will be used as the reference standard. If participants do not undergo prostate biopsy, participant follow-up (PSA level, prostate imaging, or later biopsy) will be used as reference standard
Proportion of prostate lesions determined to be cancer determined by [Ga-68]PSMA compared to histopathology | During scan, up to 35 minutes
  Quantitative data collected from PET biomarker ([Ga-68]PSMA) uptake will be used to analyze prostate lesions for differentiation between benign prostate changes and prostate cancer. Differentiation prostate lesion by PET biomarker will be compared to histology reference standard.

SECONDARY OUTCOMES:
Determination of prostate lesion aggressiveness using Gleason scores | During scan, up to 35 minutes
  Uptake of ([Ga-68]PSMA) will be compared with the Gleason score, which is a grading system used to determine the aggressiveness of prostate cancer. Scores range from 2 to 10, with higher scores indicating worse outcomes (more likely that the cancer will grow and metastasize)
Determination of prostate lesion aggressiveness using prostate grading system scores | During scan, up to 35 minutes
  Uptake of ([Ga-68]PSMA) wil be compared with the prostate grading system score, which is an extension of the current Gleason grading scale for determining the stage and aggressiveness of prostate cancer. This system is designed to provide a simplified and more accurate grading stratification system than the current Gleason Score.
  Scores range from 1 to 5, with higher scores indicating worse outcomes
Average pre-test PSA level | During scan, up to 35 minutes
  Average pre-test PSA level will be measured and reported. Ability of digital PET/CT using [Ga-68]PSMA uptake to identify malignant prostate lesions will be explored by plotting PSA levels against diagnostic performance of PET/CT using [Ga-68]PSMA, with histopathology serving as the reference standard.
Proportion of metastatic lesions identified by digital PET/CT using [Ga-68]PSMA compared to reference | During scan, up to 35 minutes
  Focally increased [Ga-68]PSMA uptake within the torso PET images will be compared with standard of care clinical imaging to verify the presence of metastatic lesions. In addition, patient follow up and histopathology will be used as reference if available.

OTHER OUTCOMES:
Optimized image reconstruction parameters - Voxel size | During scan, up to 35 minutes
  The acquired datasets from digital PET/CT using [Ga-68]PSMA will be reconstructed in different voxel sizes and by using dedicated reconstruction parameters affecting the noise levels of the images. Optimized image reconstruction parameters will be identified, including "voxel size" and "image quality"
  - Voxel size: 4x4x4mm, 2x2x2mm, 1x1x1mm
Optimized image reconstruction parameters - Image quality | During scan, up to 35 minutes
  The acquired datasets from digital PET/CT using [Ga-68]PSMA will be reconstructed in different voxel sizes and by using dedicated reconstruction parameters affecting the noise levels of the images. Optimized image reconstruction parameters will be identified, including "voxel size" and "image quality"
  - Image quality, assessed via visual analysis focused on the separation of anatomical structures (.e.g. delineation of the pelvis) and abnormal findings, e.g. increased tracer uptake within the prostate gland
Optimized acquisition and reconstruction parameters of digital PET - Image quality | During scan, up to 35 minutes
  Acquired PET/CT data sets will be reconstructed using different algorithms including respiratory and cardiac motion. The impact of variation in acquisition and reconstruction parameters on quantification of PET images will be assessed as well, Including "image quality" and "iterations and subsets"
  - Image quality, assessed via visual analysis focused on the separation of anatomical structures (.e.g. delineation of the pelvis) and abnormal findings, e.g. increased tracer uptake within the prostate glan
Optimized acquisition and reconstruction parameters of digital PET - Iterations and subsets | During scan, up to 35 minutes
  Acquired PET/CT data sets will be reconstructed using different algorithms including respiratory and cardiac motion. The impact of variation in acquisition and reconstruction parameters on quantification of PET images will be assessed as well, Including "image quality" and "iterations and subsets"
  - Iterations and subsets are part of the Iterative Reconstruction used for PET image reconstruction. Ordered subsets methods group projection data into an ordered sequence of subsets (or blocks). An iteration of ordered subsets EM is defined as a single pass through all the subsets, in each subset using the current estimate to initialize application of EM with that data subset.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Avril, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data